CLINICAL TRIAL: NCT07119008
Title: Use of Virtual Reality as a Cognitive Remediation Tool in the Depressed Elderly Subject
Brief Title: Use of Virtual Reality as a Tool for Cognitive Remediation in Elderly Depressed Patients
Acronym: REVIVED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 29BRC23.0272 - REVIVED
Record Dates: First submitted 2025-06-20; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Virtual Reality; Depression
Keywords: virtual reality
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Clinical investigation of a Class I medical device. Early interventional, uncontrolled, single-center, unblinded trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- use of virtual reality (Experimental)
  Interventions: Device: Virtual reality

INTERVENTIONS:
Device: Virtual reality — Patients will perform 12 virtual reality sessions at a rate of 2 sessions per week for 6 weeks. The patient will be offered to properly store food groceries by differentiating perishable or non-perishable foods from non-food items, or to prepare cooking recipes.

SUMMARY:
Depression, the most common mental disorder affecting the elderly, represents a major public health issue. This pathology leads to a loss of activity and autonomy in the elderly. It impairs executive skills, enabling a person to take initiatives, perform goal-oriented actions and adapt to new situations. Impaired executive functions greatly increase the risk of loss of autonomy and institutionalization, as well as the burden on caregivers. Antidepressant treatments have little or no effect on cognitive disorders. It therefore appears necessary to offer these patients specific treatment of these cognitive symptoms. The investigators are interested in cognitive remediation based on virtual reality (VR) for its ecological and modular characteristics, the innovative aspect of this technique, the appeal of virtual experiences, and their easy access to the general public. The main objective of this study is to demonstrate the acceptability of the VR technique in a population of subjects aged 70 and over, suffering from cognitive disorders and associated depression.

In this study the investigators support the use of VR as a tool for cognitive remediation and ecological staging of their interactions with caregivers in the face of executive disorders found in patients suffering from depression. By improving their cognitive skills, VR brings greater autonomy and improved quality of life for patients and their caregivers. The investigators therefore plan to use a virtual environment to create scenarios that reproduce real-life situations, which appear to be more relevant than conventional cognitive remediation exercises.

The investigators chose acceptability as the main criterion for this technique, as the elderly population is identified as a sensitive population in the opinion issued by ANSES in June 2021. What's more, this population is often excluded from the new digital technologies; it therefore seems interesting to look at the acceptability of virtual reality by this elderly population.

DETAILED DESCRIPTION:
Every patient diagnosed with depression receives psychotropic treatment comprising one or more antidepressants, possibly combined with one or more thymoregulators (e.g. bipolar patients), one or more anxiolytics and/or a hypnotic. The elderly depressive patient is also treated with supportive psychotherapy and/or group therapy at the day hospital. The trial proposes an additional tool, virtual reality, aimed at improving the cognitive abilities, particularly executive abilities, of the elderly depressive subject, thereby helping to maintain his or her functional abilities, i.e. his or her ability to stay as autonomous as possible at home and maintain a good quality of life. In fact, cognitive disorders associated with depression do not respond to antidepressant medication, if at all. It therefore seems important to optimize the treatment of depression in the elderly subject by adding a cognitive target. The investigators's project is to offer patients the opportunity to live in a virtual kitchen, where they can carry out everyday tasks. The scenario for the VR sessions has been designed in collaboration with, the principal investigator at CHU and his team, and the members of B COM and HDG involved in the study. Particular attention is paid to the fact that this scenario is intended for an elderly patient population, so as to prevent as far as possible the occurrence of cybermalaise The patient will be asked to arrange food shopping appropriately, differentiating between perishable and non-perishable foodstuffs and non-food items, or to prepare cooking recipes. Virtual reality has the advantage of being able to offer ecological, configurable activities, targeting precise tasks that call on executive functions such as initiative, anticipation and planning, mental flexibility and inhibition. Patients will undergo 12 VR sessions at a rate of 2 sessions per week for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 70 or over;
* Patient with a characterized depressive episode as assessed by the GDS (Score > 13 at inclusion);
* Patient with a minimum MMS score of 23/30 at inclusion;
* Patient affiliated to or benefiting from a social security scheme;
* Patient having received information on the protocol and having given free, informed and written consent.

Exclusion Criteria:

* Patients suffering from epilepsy;
* Patients suffering from inner ear disorders;
* Patients with balance disorders or postural instability;
* Patients with swallowing disorders requiring mixed feeding;
* Patients suffering from migraines;
* Patients with major sensory deficits (visual or auditory);
* Patients suffering from eye pathologies or abnormalities, and whose condition strictly contraindicates virtual reality;
* Patients suffering from oculo-motor disorders;
* Patients with sensory-motor deficits affecting the upper limb(s) that prevent them from performing the tasks required during VR sessions;
* Patients suffering from primary neuropathic disorders or secondary to metabolic pathologies;
* Patients suffering from acute psychiatric decompensation that makes it impossible for them to cooperate with the sessions (opposition, agitation, acute delusions, hallucinations, panic attacks);
* Patients with uncontrolled cardiac pathology (angina, heart failure, rhythm disorders, conduction disorders);
* Patients with uncontrolled hypertension (SBP > 140 mmHg and DBP > 90 mmHg in patients with traited hypertension);
* Patients with implanted medical devices (pacemakers, defibrillators, etc.);
* Patients under legal protection (guardianship) or deprived of liberty.
* Patients who do not speak or read French fluently, unable to understand the principle of the study questionnaires and unable to cooperate with the tests.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
The acceptability of Virtual Reality | at the end of session 12, on average in Week 6
  Virtual Reality acceptability will be assessed using the French version of the Acceptability E-scale questionnaire at the end of session 12. A success/failure criterion will be defined by setting the cut-off point at 24 out of 30. The questionnaire will also be completed at the end of sessions 1 and 6, to provide usable information should a patient withdraw from the protocol prematurely for any reason other than refusal to continue the study.
  A patient who decides to stop the virtual reality sessions before the 12th session will be considered as a failure.

SECONDARY OUTCOMES:
TERV tolerance | at the end of the sessions, on average in Week 6
  TERV (Virtual Reality Exposure Therapy) tolerance, which will be assessed by looking for symptoms of cybermalaise using the UQO Cybermalaise Questionnaire at the end of each session. This questionnaire includes 16 symptoms that may be experienced during the virtual reality sessions, similar to motion sickness. At the end of the sessions, the patient is asked to rate them in terms of intensity (not at all, a little, moderately, severely).
The impact of TERV on depressive symptomatology | at inclusion and at the end of the 12 sessions, on average in Week 6
  The impact of TERV on depressive symptomatology, which will be assessed using the Geriatric Depression Scale (GDS) at inclusion and at the end of the 12th session. This scale comprises 30 yes/no questions on depressive symptomatology. A score of 10 to 19 corresponds to moderate depression, and 20 to 30 to severe depression.
The impact of TERV on quality of life | at inclusion and at the end of the 12 sessions, on average in Week 6
  The impact of TERV on quality of life, which will be assessed using the Elderly Adapted Quality of Life Scale (EQVPA) at inclusion and at the end of the 12th session. This scale comprises 5 questions, each rated from 0 to 3. The score is between 0 and 15.
The impact of TERV on executive disorders | at inclusion and at the end of the 12 sessions, on average at Week 6
  The impact of TERV on executive disorders, which will be measured by a neuropsychological evaluation including: Stroop Victoria tst.
  The assessment will be carried out at inclusion and at the end of the 12th session. These tests target the executive functions of interest in this research, as depression favours the emergence of dysexecutive disorders and the loss of functional abilities in daily life.
The impact of TERV on executive disorders | At inclusion and at the end of the 12 sessions, on average at Week 6
  The impact of TERV on executive disorders, which will be measured by a neuropsychological evaluation including: WAIS IV digit memory empans test (eschler Adult Intelligence Scale)
The impact of TERV on executive disorders | At inclusion and at the end of the 12 sessions, on average at Week 6
  The impact of TERV on executive disorders, which will be measured by a neuropsychological evaluation including: Dubois test
The impact of TERV on executive disorders | At inclusion and at the end of the 12 sessions, on average at Week 6
  The impact of TERV on executive disorders, which will be measured by a neuropsychological evaluation including: BREF (Rapid Frontal Efficiency Battery) test
The impact of TERV on executive disorders | At inclusion and at the end of the 12 sessions, on average at Week 6
  The impact of TERV on executive disorders, which will be measured by a neuropsychological evaluation including: zoo test
Mental workload induced by VR sessions | at inclusion and at the end of the 12 sessions, on average at Week 6
  Mental workload induced by VR sessions, which will be measured by the NASA-TLX (NASA Task Load Index) in French at the end of each session

CONTACTS AND LOCATIONS:
Overall Officials: Sophie LE BORGNE, Dr, Principal Investigator — CHU Brest
Locations (1):
- CHU Brest - Hôpital de Bohars, Bohars, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.